CLINICAL TRIAL: NCT05030077
Title: A Single-arm, Phase II Study of Anlotinib Combined With Platinum/Gemcitabine for First Line Treatment of Advanced Urothelial Carcinoma
Brief Title: Anlotinib Combined With Platinum/Gemcitabine for First Line Treatment of Advanced Urothelial Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tianjin Medical University Second Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALTER-UC-008
Record Dates: First submitted 2021-08-16; First posted 2021-09-01 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Urothelial Carcinoma; Anlotinib; Urogenital Neoplasms; Cisplatin; Carboplatin; Gemcitabine; Antineoplastic Agents
Keywords: Urothelial Carcinoma; Chemotherapy; Anlotinib
MeSH Terms: conditions — Carcinoma, Transitional Cell; Urogenital Neoplasms | interventions — anlotinib; Cisplatin; Carboplatin; Gemcitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Anlotinib — Anlotinib(12mg) oral daily for days 1-14, 21 days per cycle
  Other Names: AL3818
Drug: Cisplatin — Cisplatin (70 mg/m2) IV day 1
Drug: Carboplatin — If the patients can't tolerate cisplatin, they will be treated with carboplatin (AUC 4.5mg/mL·min) IV day 1
Drug: Gemcitabine — Gemcitabine ( 1000 mg/m2) IV days 1 and 8

SUMMARY:
Anlotinib is a novel oral multitarget tyrosine kinase inhibitor and primary targeted to VEGFR, FGFR, PDGFR and c-Kit. This study intends to assess the efficacy and safety of anlotinib combined with platinum/gemcitabine for first line treatment of advanced urothelial carcinoma.

DETAILED DESCRIPTION:
The primary objective is to determine the antitumor activity of anlotinib combined with platinum/gemcitabine (Objective Response rate, ORR) in patients with advanced urothelial carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. 18-75 years, ECOG PS: 0-1.
2. Unresectable or metastatic urothelial carcinoma of the bladder, urethra, ureter, or renal pelvis.
3. At least one measurable lesion according to RECIST 1.1.
4. The main organ function meets the following criteria within 7 days before enrollment:

   1. Blood tests are subject to the following criteria (without blood transfusion within 14 days): hemoglobin (HB) ≥ 90g / L; neutrophil absolute value (ANC) ≥ 1.5 × 109 / L; platelets (PLT) ≥ 80 × 109 / L.
   2. Biochemical tests are subject to the following criteria: total bilirubin (TBIL) ≤ 1.5 times the upper limit of normal (ULN); alanine aminotransferase (ALT) and aspartate aminotransferase AST ≤ 2.5ULN, such as with liver metastasis, then ALT and AST ≤ 5ULN; serum creatinine (Cr) ≤ 1.5ULN or creatinine clearance (CCr) ≥ 60ml / min.
5. Women of childbearing age must have taken reliable contraceptive measures and performed a pregnancy test (serum) within 3 days prior to enrollment, and the results were negative, and were willing to use appropriate methods during the trial and 180 days after the last administration of the test drug.
6. Patients voluntarily joined the study and signed informed consent, with good adherence and follow-up.

Exclusion Criteria:

1. Pregnant or lactating women.
2. A history of hypersensitivity to the study drugs.
3. Patients have received systemic treatment.
4. Patients with uncontrolled or high-load central nervous system metastases (or with obvious symptoms)
5. Patients with other diseases, including:

   1. Hypertension and uncontrollable levels of normal anti-hypertensive medication: systolic blood pressure≥150 mmHg, diastolic blood pressure≥90 mmHg.
   2. Unstable angina, newly diagnosed with angina or acute myocardial infarction within 6 months prior to enrollment, arrhythmia ( including: QTcF of male≥450ms ) requires medical intervention congestive heart failure (New York Heart Association (NYHA)≥2)
   3. Active or uncontrollable infections (CTCAE 5.0≥2)
   4. Known history of human immunodeficiency virus infection (HIV, congenital immune deficiency disease, or a history of organ transplantation)
   5. Urinary protein ≥ ++ or 24 hours urine protein > 1 g
   6. Any malignant tumor within 5 years, except those who have been cured or stabilized.
   7. Uncured adverse events (NCI-CTCAE 5.0 grade II or greater) due to any treatment before, except for alopecia.
   8. There are many factors that affect oral drug absorption (such as inability to swallow, Postgastrointestinal resection, chronic diarrhea and intestinal obstruction, etc.).
   9. Abnormal blood coagulation (PT>16s、APTT>43s、TT>21s、Fbg<2g/L), with bleeding tendency or undergoing thrombolysis or anticoagulant therapy. Under the premise of an odds ratio (INR) ≤ 1.5, low-dose heparin (1mg daily) or low-dose aspirin (daily dose ≤ 100 mg) is allowed for preventive purposes.
   10. Patients who underwent major surgical treatment, open biopsy, or significant traumatic injury within the first 4 weeks of enrollment.
   11. Patients whose tumor has radiographically invaded an important vessel or whose tumor is determined by the investigators to be at high risk of incurring an important vessel and causing fatal hemorrhages during the study period.
   12. Patients who have seizures and need treatment.
   13. Patients with any signs of hemorrhage or history, regardless of severity; patients with any bleeding or bleeding episodes (NCI-CTCAE 5.0 grade III) within 4 weeks prior to grouping have unhealed wounds, ulcers, or fractures.
   14. Artery or venous thrombosis occurred within 6 months, such as cerebrovascular accidents (including transient ischemic attacks), deep vein thrombosis, and pulmonary embolism.
   15. Patients have been inoculated with attenuated live vaccine within 28 days before enrollment or plan to inoculate vaccine during the trial.
   16. Other systemic diseases that can't be controlled (such as diabetes, etc.).
6. Patients with other serious physical or mental illness or laboratory abnormalities that may increase the risk of participating in the study or interfere with the results of the study, as well as patients that the investigator considers unfit to participate in the study.
7. Patients who have participated in clinical trials of other antitumor drugs within four weeks.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | From date of enrollment until disease progression,assessed up to 1 year
  The objective response rate is defined as the percentage of participants with measurable lesions achieving a Complete Response (CR) or Partial Response (PR) based on Response Evaluation Criteria In Solid Tumors Version 1.1(RECIST v1.1) criteria. Per RECIST v1.1) for target lesions and assessed by MRI or CT: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), greater than or equal to (>=) 30 percent (%) decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.

SECONDARY OUTCOMES:
Duration of Response (DoR) | From date of enrollment until disease progression,assessed up to 3 years
  The duration of response (CR or PR) is defined as the earliest date a participant achieved a CR or a PR, calculated from the date of initial documentation of a response to the date of first documented evidence of progressive disease (or relapse for participants who experience CR during the study) or death.
Progression free survival (PFS) | From date of enrollment until the date of first documented progression,assessed up to 3 years
  Progression-free survival estimated using Kaplan-Meier methods is defined as the time from the date of informed consent to the earlier of death or disease progression. Patients alive without disease progression are censored at the date of last disease evaluation. Progressive disease (PD) based on RECIST 1.1 is at least a 20% increase in the sum of longest diameter (LD) of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. Equivocal progression of non-target lesions also qualifies as PD.
Overall Survival (OS) | From date of enrollment until death,assessed up to 5 years
  Overall survival is defined as the time interval in days between the date of the first dose of study drug and the participant's death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Yuanjie Niu, MD,PhD, Principal Investigator — Tianjin Medical Unversity Second Hospital
Locations (1):
- Tianjin Medical Unversity Second Hospital, Tianjin, China